CLINICAL TRIAL: NCT01646138
Title: Influenza A 2009 H1N1 Human Challenge Study in Healthy Adult Volunteers
Brief Title: Influenza A 2009 H1N1 Challenge Study in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 120077; 12-I-0077 (Other: NIH - National Institute of Allergy and Infectious Diseases)
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: H1N1; Influenza; Human; Challenge Study; Healthy Volunteer
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Challenge Virus (Experimental): The Ca/04/2009/H1N1 Vero Grown Challenge Virus was administered intranasally to each participant using a nasal sprayer. A total volume of up to 1 mL of virus will be administered.
  Interventions: Biological: Ca/04/2009/H1N1 Vero Grown Challenge Virus

INTERVENTIONS:
Biological: Ca/04/2009/H1N1 Vero Grown Challenge Virus — The human challenge virus will be administered intranasally to each participant using a nasal sprayer. A total volume of up to 1 mL of virus will be administered.

SUMMARY:
Background:

- A challenge study exposes a person to a disease and allows researchers to study the disease through the body's healing process. An influenza challenge study that looks at different amounts of the flu virus can provide more information on the smallest amount needed to cause an infection. Researchers want to give one dose of the Influenza A H1N1 virus to healthy volunteers to see how the body responds to the virus.

Objectives:

* To find the smallest dose of Influenza A H1N1 virus that may cause a mild to moderate flu infection in a healthy adult.
* To study how the body s immune system responds to the virus.

Eligibility:

* Healthy volunteers at least 18 years of age.
* Participants must be willing to remain in isolation for a minimum of 9 days.

Design:

* Participants will be admitted to a hospital inpatient isolation unit. They will be screened with a physical exam and medical history. They will also have heart and lung function tests. Blood, urine, and nasal swab/wash samples will be collected.
* Participants will receive a single nasal spray of the flu virus. They will stay on the inpatient unit for at least 9 days.
* Participants will be monitored for the length of their stay. They will have frequent blood tests and other procedures as needed.
* Participants will be allowed to go home once they have had two negative tests for the virus. The tests will be given on two consecutive days....

DETAILED DESCRIPTION:
The high morbidity and mortality associated with both pandemic and seasonal influenza, and the anticipation of future influenza pandemics, puts influenza front and center in infectious disease research. Because the natural history and pathogenesis of human influenza has not been well characterized and cannot be adequately studied in animal models or with current in vitro techniques, important questions about influenza pathogenesis can only be approached through human challenge studies.

Previous human challenge studies have addressed some aspects of the natural history of influenza by evaluating the timing of viral replication, shedding, clinical symptoms, and innate and adaptive immune responses. Although these studies have provided important information, in the United States, all but 1 were performed prior to 1990. Without exception, these studies had limitations due to the scope of the study and/or the scientific techniques available at that time.

The primary objective of this study is to determine the dose of influenza A 2009 H1N1 human challenge virus that will induce a mild to moderate uncomplicated influenza infection in healthy volunteers. This protocol will examine some of the basic questions that remain unanswered regarding the pathogenesis of influenza in humans, namely, a detailed clinical and immunological characterization of uncomplicated influenza viral pathogenesis in healthy adult volunteers.

Secondary objectives will evaluate clinical disease, length of viral shedding, and pathogenesis in those with influenza infection including identification of clinical markers of the disease. Notably, the exploratory objectives will seek to discover viral factors necessary for human infection/adaptation and to evaluate host immune response, viral replication, viral fitness, and the intrahost evolution.

Collaboration between National Institute of Allergy and Infectious Diseases (NIAID) investigators and outside scientists will generate opportunities to further develop and expand areas of clinical influenza research based on the proposed challenge model.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Greater than or equal to 18 and less than or equal to 50 years of age.
2. Agrees to not use tobacco products during participation in this study.
3. Willingness to remain in isolation for the duration of viral shedding (at a minimum 9 days) and to comply with all study requirements.
4. A female participant is eligible for this study if she is not pregnant or breast feeding and 1 of the following:

   * Of non-childbearing potential (i.e., women who have had a hysterectomy or tubal ligation or are postmenopausal, as defined by no menses in greater than or equal to 1 year).
   * Of childbearing potential but agrees to practice effective contraception or abstinence for 4 weeks prior to and 8 weeks after administration of the influenza challenge virus. Acceptable methods of contraception include 1 or more of the following: 1) male partner who is sterile prior to the female participant s entry into the study and is the sole sexual partner for the female participant; 2) implants of levonorgestrel; 3) injectable progestogen; 4) an intrauterine device with a documented failure rate of < 1%; 5) oral contraceptives; and 6) double barrier methods including diaphragm or condom with a spermicide.
5. Willing to have samples stored for future research.
6. Prechallenge serum hemagglutination-inhibition titer against the challenge strain of 1:16 or less.
7. HIV uninfected.

EXCLUSION CRITERIA:

1. Presence of self-reported or medically documented significant medical condition including but not limited to:

   1. Chronic pulmonary disease (e.g., asthma, emphysema).
   2. Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
   3. Chronic medical conditions requiring close medical follow-up or hospitalization during the past 5 years (e.g., diabetes mellitus, renal dysfunction, hemoglobinopathies).
   4. Immunosuppression or ongoing malignancy.
   5. Neurological and neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
   6. Postinfectious or postvaccine neurological sequelae.
2. Have close or household (i.e., share the same apartment or house) high-risk contacts including but not limited to:

   1. Persons greater than or equal to 65 years of age.
   2. Children < 5 years of age.
   3. Residents of nursing homes.
   4. Persons of any age with significant chronic medical conditions such as:

      * Chronic pulmonary disease (e.g., asthma).
      * Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
      * Contacts who required medical follow-up or hospitalization during the past 5 years because of chronic metabolic disease (e.g., diabetes mellitus, renal dysfunction, hemoglobinopathies).
      * Immunosuppression or cancer.
      * Neurological and neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
      * Children and teenagers who are receiving long-term aspirin therapy.
      * Women who are pregnant or who are trying to become pregnant.
3. Individual with body mass index (BMI) less than or equal to 18.5 and greater than or equal to 40.
4. Smokes more than 4 cigarettes or other tobacco products on weekly basis.
5. Complete blood count (CBC) with differential outside of the NIH Department of Laboratory Medicine (DLM) normal reference range and deemed clinically significant by the PI.
6. Chemistries in the acute care, mineral, and/or hepatic panels, and/or any of the following: lactate dehydrogenase, uric acid, creatine kinase, and total protein outside of the NIH DLM normal reference range and deemed clinically significant by the PI.
7. Urinalysis outside of the NIH DLM normal reference range and deemed clinically significant by the PI.
8. Clinically significant abnormality on electrocardiogram .
9. Clinically significant abnormality as deemed by the PI on echocardiographic testing.
10. Recent acute illness within 1 week of admission to the isolation facility.
11. Known allergy to treatments for influenza (including but not limited to oseltamivir, nonsteroidals).
12. Known allergy to 2 or more classes of antibiotics (e.g., penicillins, cephalosporins, fluoroquinolones, or glycopeptides).
13. Receipt of blood or blood products (including immunoglobulins) within 3 months prior to enrollment.
14. Receipt of any unlicensed drug within 3 months or 5.5 half lives (whichever is greater) prior to enrollment.
15. Receipt of any unlicensed vaccine within 6 months prior to enrollment.
16. Self-reported or known history of current alcoholism or drug abuse, or positive urine/serum test for drugs of abuse (i.e., amphetamines, cocaine, benzodiazepines, opiates, or metabolites, but not tetrahydrocannabinol(THC) or metabolites).
17. Self-reported or known history of psychiatric or psychological issues deemed by the PI to be a contraindication to protocol participation
18. Known close contact with anyone known to have influenza in the past 7 days.
19. Any condition that, in the judgment of the Principal Investigator, is a contraindication to protocol participation or impairs the volunteer s ability to give informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Memoli, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through the NIH data repository BTRIS - Biomedical Translational Research Information System

REFERENCES:
- [Background] Hayden FG, Fritz R, Lobo MC, Alvord W, Strober W, Straus SE. Local and systemic cytokine responses during experimental human influenza A virus infection. Relation to symptom formation and host defense. J Clin Invest. 1998 Feb 1;101(3):643-9. doi: 10.1172/JCI1355. PMID 9449698
- [Background] Jameson J, Cruz J, Ennis FA. Human cytotoxic T-lymphocyte repertoire to influenza A viruses. J Virol. 1998 Nov;72(11):8682-9. doi: 10.1128/JVI.72.11.8682-8689.1998. PMID 9765409
- [Background] McAuley JL, Hornung F, Boyd KL, Smith AM, McKeon R, Bennink J, Yewdell JW, McCullers JA. Expression of the 1918 influenza A virus PB1-F2 enhances the pathogenesis of viral and secondary bacterial pneumonia. Cell Host Microbe. 2007 Oct 11;2(4):240-9. doi: 10.1016/j.chom.2007.09.001. PMID 18005742
- [Derived] Memoli MJ, Han A, Walters KA, Czajkowski L, Reed S, Athota R, Angela Rosas L, Cervantes-Medina A, Park JK, Morens DM, Kash JC, Taubenberger JK. Influenza A Reinfection in Sequential Human Challenge: Implications for Protective Immunity and "Universal" Vaccine Development. Clin Infect Dis. 2020 Feb 14;70(5):748-753. doi: 10.1093/cid/ciz281. PMID 30953061
- [Derived] Memoli MJ, Czajkowski L, Reed S, Athota R, Bristol T, Proudfoot K, Fargis S, Stein M, Dunfee RL, Shaw PA, Davey RT, Taubenberger JK. Validation of the wild-type influenza A human challenge model H1N1pdMIST: an A(H1N1)pdm09 dose-finding investigational new drug study. Clin Infect Dis. 2015 Mar 1;60(5):693-702. doi: 10.1093/cid/ciu924. Epub 2014 Nov 20. PMID 25416753
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-I-0077.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 49 participants were enrolled but 1 participant did not receive the intervention.
Groups:
- 10^3 TCID 50: Participants received Ca/04/2009/H1N1 Vero Grown Challenge Virus at a dose of 10^3 TCID50 in 1ml given intranasally.
- 10^4 TCID 50: Participants received Ca/04/2009/H1N1 Vero Grown Challenge Virus at a dose of 10^4 TCID50 in 1ml given intranasally.
- 10^5 TCID 50: Participants received Ca/04/2009/H1N1 Vero Grown Challenge Virus at a dose of 10^5 TCID50 in 1ml given intranasally.
- 10^6 TCID 50: Participants received Ca/04/2009/H1N1 Vero Grown Challenge Virus at a dose of 10^6 TCID50 in 1ml given intranasally.
- 10^7 TCID 50: Participants received Ca/04/2009/H1N1 Vero Grown Challenge Virus at a dose of 10^7 TCID50 in 1ml given intranasally.
Period: Overall Study
Arm/Group | 10^3 TCID 50 | 10^4 TCID 50 | 10^5 TCID 50 | 10^6 TCID 50 | 10^7 TCID 50
Started | 5 | 4 | 5 | 19 | 15
Completed | 5 | 4 | 5 | 19 | 13
Not Completed | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- 10^4 TCID 50: Participants received influenza A(H1N1) pdm09 at a dose of 10^4 TCID50 administered intranasally.
- 10^5 TCID 50: Participants received influenza A(H1N1) pdm09 at a dose of 10^5 TCID50 administered intranasally.
- 10^6 TCID 50: Participants received influenza A(H1N1) pdm09 at a dose of 10^6 TCID50 administered intranasally.
- 10^7 TCID 50: Participants received influenza A(H1N1) pdm09 at a dose of 10^7 TCID50 administered intranasally.
- Total: Total of all reporting groups
Arm/Group | 10^3 TCID 50 | 10^4 TCID 50 | 10^5 TCID 50 | 10^6 TCID 50 | 10^7 TCID 50 | Total
Number analyzed (Participants) | 5 | 4 | 5 | 20 | 15 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 5 | 20 | 15 | 49
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 3 | 9 | 5 | 19
  Male | 3 | 4 | 2 | 11 | 10 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 5 | 4 | 5 | 18 | 14 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 3 | 11 | 7 | 26
  White | 3 | 1 | 2 | 6 | 7 | 19
  More than one race | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent MMID
Description: Percent of individuals experiencing mild to moderate influenza infection (MMID, defined as active shedding and symptoms of influenza A) in each dosing group.
Time Frame: 67 days after influenza inoculation
Population: Analysis of the subjects who completed the study after receiving a particular dose of Ca/04/2009/H1N1 Vero Grown Challenge Virus.
Measure: Number; unit: percentage of participants
Groups:
- 10^3 TCID 50: Participants received influenza A(H1N1) pdm09 at a dose of 10^3 TCID 50 administered intranasally.
Arm/Group | 10^3 TCID 50 | 10^4 TCID 50 | 10^5 TCID 50 | 10^6 TCID 50 | 10^7 TCID 50
Number analyzed (Participants) | 5 | 4 | 5 | 19 | 13
percentage of participants | 0 | 0 | 20 | 47 | 69

ADVERSE EVENTS:
Arm/Group | 10^3 TCID 50 | 10^4 TCID 50 | 10^5 TCID 50 | 10^6 TCID 50 | 10^7 TCID 50
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/5 | 0/19 | 0/15
Other Adverse Events (participants affected / at risk) | 1/5 | 1/4 | 0/5 | 8/19 | 7/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10^3 TCID 50 (N=5) | 10^4 TCID 50 (N=4) | 10^5 TCID 50 (N=5) | 10^6 TCID 50 (N=19) | 10^7 TCID 50 (N=15)
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase (Investigations) | 0 | 1 | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 2 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes